CLINICAL TRIAL: NCT02695121
Title: Comparison of the Risk of Cancer Between Patients With Type 2 Diabetes Exposed to Dapagliflozin and Those Exposed to Other Antidiabetic Treatments
Brief Title: Cancer in Patients on Dapagliflozin and Other Antidiabetic Treatment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00007; EUPAS12116 (Registry Identifier: ENCePP)
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Bladder Cancer
MeSH Terms: conditions — Breast Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Female breast cancer: females with type 2 diabetes who are new users of dapagliflozin and females who are new users of antidiabetic drugs (ADs) in classes other than sodium-glucose cotransporter 2 (SGLT2) inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy
- Sex combined bladder cancer: male and female patients with type 2 diabetes who are new users of dapagliflozin and those who are new users of ADs in classes other than SGLT2 inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy
- Male bladder cancer: male patients with type 2 diabetes who are new users of dapagliflozin and those who are new users of ADs in classes other than SGLT2 inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy
- Female bladder cancer: female patients with type 2 diabetes who are new users of dapagliflozin and those who are new users of ADs in classes other than SGLT2 inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy

SUMMARY:
The primary objectives of this study are (1) to compare the incidence of breast cancer, by insulin use at cohort entry, among females with type 2 diabetes who are new users of dapagliflozin and females who are new users of antidiabetic drugs (ADs) in classes other than sodium-glucose cotransporter 2 (SGLT2) inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy and (2) to compare the incidence of bladder cancer, by insulin use at the index date and by pioglitazone use at the index date, among male and female patients with type 2 diabetes who are new users of dapagliflozin and those who are new users of ADs in classes other than SGLT2 inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy. Secondary objectives will compare, by insulin use at cohort entry, frequency of several measures of health care use, baseline characteristics, and incidence of selected other cancers in males and females between the two exposure cohorts.

DETAILED DESCRIPTION:
This is a multinational cohort database study to estimate the incidence of female breast cancer and bladder cancer, by insulin use at cohort entry, in patients who are prescribed dapagliflozin compared to patients prescribed other specific oral antidiabetic drugs. Dapagliflozin and other antidiabetic drugs are used to treat type 2 diabetes mellitus. Because of the mechanism of action for dapagliflozin and results from small safety monitoring studies, there is interest in further evaluating the safety of dapagliflozin in a large populations.

The study will be implemented in four administrative health care data sources in three countries: in the United Kingdom, the Clinical Practice Research Datalink (CPRD); in the United States, the Centers for Medicare and Medicaid Services (CMS) Medicare databases and the HealthCore Integrated Research Database (HIRDSM); and, in the Netherlands, the PHARMO Database Network. Individuals in the databases will be included in the study if they meet the following age criteria; 40 years or older (CPRD and PHARMO), 40 to 64 years (HIRD) or 65 years or older (Medicare); and if they did not have type 1 diabetes, were treated with one of the study drugs and meet the criteria of at least 180 days of electronic data before their first prescription of the study drug. The study period starts November 13, 2012 in CPRD, November 1, 2013 in PHARMO and January 9, 2014 in the United States data sources, and will end at the latest available data at each database at the time of analysis

ELIGIBILITY:
Inclusion Criteria:

1. patient was newly prescribed dapagliflozin or newly prescribed an AD (with or without other ADs) in a class other than SGLT2 inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy on the prescription index date
2. patient is aged 40 years or older at cohort entry; and
3. patient was enrolled in the data source for at least 180 days before the prescription index date.

Exclusion Criteria:

1. any evidence of diagnosis of type 1 diabetes before cohort entry or use of insulin alone as the first recorded AD;
2. any diagnosis of cancer before cohort entry (other than nonmelanoma skin cancer);
3. any recording of hematuria before cohort entry;
4. any cystoscopy or urine cytology performed before cohort entry;
5. any breast biopsy performed before cohort entry.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients must meet all of the inclusion criteria and none of the exclusion criteria. Comparator patients will be randomly selected in a 4:1 ratio to the dapagliflozin patients.
Sampling Method: Non-Probability Sample
Enrollment: 2133575 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of breast cancer | Index day up to twelve years
  Patients will be followed from their index date (date of first study drug prescription or dispensing) until the earliest of occurrence of one of the following: first occurrence of any one of the study endpoints, death, addition of a non-dapagliflozin SGLT2 inhibitor, disenrollment from the study database or transfer out of the GP practice, or end of the study period up to twelve years.
Incidence of bladder cancer | Index day up to twelve years
  Patients will be followed from their index date (date of first study drug prescription or dispensing) until the earliest of occurrence of one of the following: first occurrence of any one of the study endpoints, death, addition of a non-dapagliflozin SGLT2 inhibitor, disenrollment from the study database or transfer out of the GP practice, or end of the study period up to twelve years.

SECONDARY OUTCOMES:
Incidence of compsite cancer outcomes | Index day up to twelve years
  Patients will be followed from their index date (date of first study drug prescription or dispensing) until the earliest of occurrence of one of the following: first occurrence of any one of the study endpoints, death, addition of a non-dapagliflozin SGLT2 inhibitor, disenrollment from the study database or transfer out of the GP practice, or end of the study period up to twelve years.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Gutierrez, Principal Investigator — RTI Health Solutions
Locations (4):
- United States (2):
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
- Research Site, Utrecht, Netherlands
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at http://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at http://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home